CLINICAL TRIAL: NCT06309680
Title: Accuracy of Metagenomic Blood Sampling to Identify Pathogen in Infective Endocarditis Patients
Acronym: AMetIP
Status: Active, not recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other); Quadram Institute Bioscience (Other)
Responsible Party: Sponsor
Other Study IDs: 280992
Record Dates: First submitted 2024-02-09; First posted 2024-03-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Infective Endocarditis
Keywords: endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. EDTA peripheral blood sample
  2. Heart Valve tissue sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infective Endocarditis is an infection, usually a bacterium, which attacks the heart and can cause valves to leak and produces a bacterial mass which can break off from the valves and block the blood supply to important organs.

We are very keen to improve the treatment of this disease and we are measuring the impact of the treatments that we give to patients so that we have a very clear idea of which treatments work best and also which treatments are less successful.

A key part of the treatment is the accurate determination of the causative organism which allows appropriate targeted antibiotic and antifungal medication to be administered.

Accurate antibiotic regimes require detection of the causative organism and its sensitivities to each antibiotic. Antibiotic choice is then based on effectiveness, toxicity, ease of use and national guidelines. The current best technique for identifying bacteria is blood culture where organisms are identified by growing them from blood samples. However, this takes up to 5 days from sampling, resulting in delays to the correct diagnosis. Until this time, treatment requires the use of generic, more toxic antibiotic regimes.

New techniques are emerging to identify causative organisms from blood. Metagenomics allows the sequencing of bacterial DNA allowing precise identification of the infecting organism.

DETAILED DESCRIPTION:
Infective Endocarditis (IE) occurs when bacteria or fungi settle on heart valves and damage the tissues. The disease can be catastrophic and result in death, heart failure, stroke, kidney failure and other complications. Valvular damage requires cardiac surgery in approximately 50% with endocarditis; early antibiotic treatment reduces complications and improves prognosis, reducing the need for surgery. This is dependent on rapid, accurate determination of the causative organism to administer effective and targeted antimicrobial therapy.

The current best technique for identifying bacteria is blood culture - organisms are identified by growing them from blood. However, this typically takes up to 5 days.

In up to 18% of patients, blood culture fails to identify a causative organism - Blood Culture Negative Infective Endocarditis (BCNIE). As a result, patients are treated with broader spectrum antibiotics which have greater toxicity than targeted regimens, resulting in higher complication rates. Alternative technologies to standard blood culture are therefore needed.

Clinical metagenomics (CMg) allows the sequencing of bacterial DNA from blood samples allowing precise, rapid identification of the pathogen. Hitherto, this technology was expensive and limited. New technology is changing the face of CMg and will potentially allow organisms to be rapidly identified at low cost.

Barts Heart Centre (BHC) is one of the largest cardiac centres in the world, managing 150 IE cases annually. Whilst mortality for IE remains high - 17.1% in the recently published EuroENDO study - in hospital mortality at Barts Heart Centre is ~13%.

The Quadram Institute (QI) is a Biotechnology and Biological Sciences Research Council (BBSRC) funded research institute has special expertise in CMg, including two Nature papers.

This study of 200 patients will assess the accuracy of blood CMg and identify the best time to sample along with its cost effectiveness. Patients will be asked for an extra 10 mL of blood which will be sent to QI along with a routinely taken admission blood sample.

In addition if surgery is clinically required, some of the resected heart valve tissue will also be sent for CMg analysis Results from CMg will be compared to blood culture. A control group of patients undergoing valve surgery for non-IE indications will also be recruited.

To assist future commissioning of a clinical CMg service within the NHS, a cost-effectiveness analysis of use of CMg in the endocarditis diagnosis and treatment pathway will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with possible or confirmed IE referred to BHC Endocarditis MDT
* Age >18
* Able and willing to give informed consent

Exclusion Criteria:

* Patients whose diagnosis of endocarditis is "rejected" by the MDT. If this occurs after entry to the study samples will be discarded and the patient informed.
* Patients who have been treated with intravenous antibiotics for more than 7 days at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample will be a consecutive group of patients from hospitals in the trial referred to BHC Endocarditis MDT meeting for management of their disease. Approximately 150 cases are referred to the Endocarditis MDT each year and we reject the diagnosis of endocarditis in 17% of patients by the time of discharge (the cases are highly selected by the time they are referred).
  The study is designed to be practicable and applicable to a real-world group of patients. Thus, we will study all patients who give consent and have possible or definite endocarditis as per the determination of the clinical Endocarditis MDT. In practice, by the time treatment is completed the number left in the possible endocarditis group is very small (<5%) although when the patient is first referred approximately 20% are in that category. As the disease progresses down its course, the correct diagnosis quickly becomes apparent - especially after surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of CMg in blood | 3 years
  The primary objective of this study is to compare the organisms found from metagenomic testing of blood samples with organisms found from blood culture from a prospective series of sequential patients with IE and compared to blood culture, surgically-resected valve tissue culture (where surgery is undertaken) and opinion of a clinical reference group

SECONDARY OUTCOMES:
To evaluate the results of Nanopore CMg in identifying the causative organism in patients with BCNIE | 3 years
  Any organism identified will be graded by an expert panel into one of three categories:
  1. Blood culture negative, Nanopore CMg negative
  2. Blood culture negative, CMg positive, Organism unlikely to cause IE
  3. Blood culture negative, CMg positive, Organism likely to cause endocarditis We will also send tissue samples for nanopore CMg from all patients operated upon. The identification of the same organism from blood and valve tissue (taken on separate occasions) almost certainly indicates that IE was caused by the organism
1. Optimal timing of blood sampling | 3 years
  The optimal timing of blood sampling for nanopore CMg in IE is unknown. Thus, we will examine the first available Ethylenediaminetetraacetic acid (EDTA) stored sample retained in the labs nd compare it to the results of a sample taken especially for the study, probably a few days later.
3. Metagenomic Techniques | 3 years
  We will compare two different metagenomic techniques - 16s blood testing and host suppression on Nanopore platform.

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital. West Smithfield, London, United Kingdom